CLINICAL TRIAL: NCT05209594
Title: Evaluation of the Healthy Relationships Program for 2SLGBTQIA+ Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113468
Record Dates: First submitted 2021-10-03; First posted 2022-01-26 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Adolescent Development
Keywords: Mental health; Social emotional functioning; Gender identity; Sexual identity
MeSH Terms: conditions — Psychological Well-Being | interventions — Horseradish Peroxidase

STUDY DESIGN:
Intervention Model Description: GSA members (students in grades 9 to 12) will be assessed in one of two arms. The intervention arm includes GSAs that will implement the Healthy Relationships Program (HRP) for two-spirit, lesbian, gay, bisexual, trans, queer, intersex, and asexual (2SLGBTQIA+) youth. The comparison arm will be GSAs where standard GSA programming is delivered.
Masking Description: Due to the nature of the intervention, it is not possible to have blinded conditions. Most school-based prevention programs of this type are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Relationships Program (HRP) for 2SLGBTQIA+ Youth (Experimental): Students in grades 9 to 12 participating in GSAs where the HRP for 2SLGBTQIA+ Youth is being implemented.
  Interventions: Behavioral: Healthy Relationships Program (HRP) for 2SLGBTQIA+ Youth
- Regular GSA Programming (Active Comparator): Students in grades 9 to 12 participating in regular GSA programming.
  Interventions: Behavioral: Standard GSA Programming

INTERVENTIONS:
Behavioral: Healthy Relationships Program (HRP) for 2SLGBTQIA+ Youth — The Healthy Relationships Program (HRP) for Two-Spirit, Lesbian, Gay, Bisexual, Trans, Queer, Intersex, and Asexual + (2SLGBTQIA+) Youth is a small group positive mental health promotion program for gender, sexual, and romantic minority youth. It helps build resiliency and promote well-being among 2SLGBTQIA+ youth. It affirms, validates, and celebrates sexual and gender diversity, cultivates a caring and supportive community, and helps 2SLGBTQIA+ youth develop skills and strategies that promote healthy relationships. This trauma-informed, strengths-focused program explores stressors unique to 2SLGBTQIA+ youth, including identity and expression invalidation, stigma, prejudice and discrimination, internalized oppression, coming out, safety, and microaggressions. This program includes 17 sessions, each lasting approximately 45 minutes. It may be delivered in school-based Genders and Sexualities Alliances/Gay-Straight Alliances (GSA) or 2SLGBTQIA+ youth group settings.
  Arms: Healthy Relationships Program (HRP) for 2SLGBTQIA+ Youth
Behavioral: Standard GSA Programming — Students at comparison sites will participate in standard GSA programming, a safe space for 2SLGBTQIA+ youth and their allies to meet, develop relationships, support each other, socialize, and learn about sexuality and gender-related topics, and lobby for social change.
  Arms: Regular GSA Programming

SUMMARY:
The Healthy Relationships Program (HRP) for two-spirit, lesbian, gay, bisexual, trans, queer, intersex, and asexual (2SLGBTQIA+) Youth is a flexible and adaptable 17-session mental health promotion and healthy relationship program for gender, sexual, and romantic minority youth. It helps build resiliency and promote well-being among 2SLGBTQIA+ youth. It affirms, validates, and celebrates sexual and gender diversity, cultivates a caring and supportive community, and helps 2SLGBTQIA+ youth develop skills and strategies that promote healthy relationships. Investigators will evaluate the HRP for 2SLGBTQIA+ youth in 10 intervention and 10 comparison Genders and Sexualities Alliance/Gay-Straight Alliances (GSAs) in schools across Canada. GSA advisors (educators) at intervention schools will receive training in the program prior to implementation. GSA members (students in grades 9 to 12) at both intervention and comparison sites will participate in a survey at three time points: (1) pre-GSA programming survey at the beginning of the school year, (2) a post-GSA programming survey at the end of the school year, and (3) a follow-up survey at the beginning of the next school year. The primary outcome is social-emotional functioning.

DETAILED DESCRIPTION:
Study Background and Design:

Two-spirit, lesbian, gay, bisexual, trans, queer, intersex, and asexual (2SLGBTQIA+) youth experience disproportionately negative outcomes compared to their heterosexual and cisgender peers in a range of domains, including mental health, problematic substance use, and violence. The heightened risk experienced by these youth appears to be in large part a function of the discrimination and minority stress that they face. Antihomophobic and anti-transphobic school policies and programs can play a protective role in the lives of 2SLGBTQIA+ youth. For example, 2SLGBTQIA+ youth who attend schools that have Genders and Sexualities Alliance/Gay-Straight Alliances (GSAs) are at a lower risk for negative health behaviours, including alcohol and substance use and report increased psychological well-being and psychosocial functioning. Research has found that school staff (e.g., GSA advisors) require more guidance, training, networking opportunities to build their capacity to support 2SLGBTQIA+ youth. Some prominent program developers/academics in the field have suggested that GSAs should offer structured programming depending on the needs and desired of each group, to encourage 2SLGBTQIA+ youth to process and cope with victimization in healthy ways.

The Healthy Relationships Program (HRP) for 2SLGBTQIA + Youth fills a gap in mental health promotion and healthy relationship programming for queer, trans, and gender diverse youth. The program has been piloted in Ontario schools and community agencies and was well received by both facilitators and participants. This study will scale up our previous work and undertake a quasi-experimental, mixed-method evaluation of the HRP for 2SLGBTQIA+ youth with school partners across Canada. The HRP for 2SLGBTQIA+ Youth will be delivered nationally within 10 high school GSAs, and 10 GSAs with standard programming will be utilized as a comparison group. GSA members (students in grades 9 to 12) will participate in pre, post and follow-up surveys. The use of three-time points allows the investigators to look at program impacts within a reasonable timeframe, and to identify potential mechanisms at post-intervention that could mediate changes at follow-up.

By comparing the experiences of GSA members who participate in the HRP for 2SLGBTQIA+ Youth with those who participate in standard GSA programming, investigators will be able to evaluate the relative benefits of standard GSA programming versus formalized/structured programming. Specifically, investigators will be able to determine the extent to which the HRP for 2SLGBTQIA+ Youth promotes positive mental health and well-being among 2SLGBTQIA+ youth and their allies. The study will identify changes in social-emotional assets and resilience, youth well-being, mental health, identity affirmation, dating violence and help-seeking.

Participants:

GSA members (students in grades 9 to 12) participating in high school GSAs where the HRP for 2SLGBTQIA+ Youth is delivered, and GSA members participating in high school GSAs delivering standard programming. Although GSAs vary in size, investigators conservatively estimate that approximately 100 GSA members will participate in this study (i.e., 5 youth from each of the 20 schools - 10 intervention and 10 non-intervention). However, the total number of youth participants may vary considerably since GSAs vary in size (2 to 30+ students).

Procedures:

The school boards partnering on this study will assist in identifying intervention and comparison school sites within their district. All intervention GSA advisors will receive a two-day training on the HRP for 2SLGBTQIA+ youth. GSA members (students in grades 9 to 12) from intervention and comparison sites will be invited to participate in any of the following research activities:

1. A pre-GSA programming survey at the beginning of the school year (October/November 2021).
2. A post-GSA programming survey at the end of the school year (May/June 2022).
3. A follow-up survey at the beginning of the next school year (October 2022). They will also be invited to participate in an interview at the end of the school year.

Investigators will recruit a second cohort the following year if needed to reach the sample size (i.e., number of schools). If a second cohort is included, the timing would be:

A pre-GSA programming survey at the beginning of the school year (October/November 2022).

2. A post-GSA programming survey at the end of the school year (May/June 2023). 3. A follow-up survey at the beginning of the next school year (October 2023). They will also be invited to participate in an interview at the end of the school year.

GSA members will consent to their own participation to protect them for requiring to disclose their sexual orientation and/or gender identity to their parents as a condition for research participation. Guardian consent will only be obtained if absolutely required by a partnering school board.

Planned analyses:

Investigators will explore the pre-test data through bivariate analyses to investigate baseline equivalency between intervention and comparison groups using chi-square or t-test as appropriate; any unbalanced covariates will be controlled for in multivariate models. (If two cohorts, cohort differences on baseline characteristics will also be investigated). Youth will be clustered within GSAs, and so associations with outcomes variables at follow-up will be explored using multilevel models. This will allow us to control for both individual and site-level covariates. Intent-to-test analyses will be used, and missing data will be addressed using full information maximum likelihood. The main predictor for all models will be group status (intervention vs. comparison).

ELIGIBILITY:
Inclusion Criteria:

* All students participating in the GSA at invention and comparison sites are eligible to participate
* Age 13 to 19 years old

Exclusion Criteria:

* Students with low literacy or cognitive functioning may not be able to complete the self-report measures.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Positive social-emotional functioning | Change from baseline to four month follow-up (up to 12 months)
  Measured by the Social-Emotional Assets and Resiliency Scales-Adolescent (SEARS-A) that assesses social-emotional assets of responsibility, self-regulation, social competence, and empathy. Participants respond to the 35 items on a 4-point Likert scale (0 = never, 1 = sometimes, 2 = often, 3 = always). The combined total score ranges from 0 to 105 with higher scores indicating greater social-emotional strengths.

SECONDARY OUTCOMES:
Gender Sexuality Alliance (GSA) functioning | Change from baseline to four month follow-up (up to 12 months)
  GSA functioning as measured by the adapted school climate and connectedness survey. Participants respond to the 39 items on a 5-point Likert scale from strongly disagree to strongly agree. The total score ranges from 39 to 195.
Dating violence | Change from baseline to four month follow-up (up to 12 months)
  Dating violence perpetration as measured by the Conflict in Adolescent Dating Relationships Inventory (short form). Participants respond to the 20 items on a 4-point Likert scale (0 = never, 1 = seldom, 2 = sometimes, 3 = often). The sum of the perpetrator and victimization items are calculated (10 items each). Scores range from 0 to 30 with higher scores indicating a higher incidence of abusive behaviour (perpetrator items) or victim of abuse (victimization items).
Help-seeking intentions | Change from baseline to four month follow-up (up to 12 months)
  Self-reported intentions to seek help as measured by General Help-seeking Questionnaire. Participants indicate their likelihood to seek help for a personal or emotional problem from the people listed on a 4-point Likert scale (1= very unlikely, 2=unlikely, 3=likely, 4=very likely). A mean score is calculated on the items with the higher score indicating a higher likelihood to seek help for a problem.
Actual help-seeking | Change from baseline to four month follow-up (up to 12 months)
  Actual help-seeking over the past 2 weeks as measured by the Actual Help Seeking Questionnaire. Participants check the people they have sought help from over a two-week period for a personal or emotional problem and then describe the type of problem. A score for the total number of people they sought help from is calculated and open-ended descriptions are coded for type of problem (e.g., mental health, relationships, school, etc.).
Positive mental health | Change from baseline to four month follow-up (up to 12 months)
  Emotional well-being and aspects of psychological and social functioning that occur within the past month as measured by the Adolescent Mental Health Continuum-Short Form. Participants rate 14 items on a 6-point Likert scale from 0=Never to 5 = Every day. Scores range from 0 to 70 with higher scores indicating higher experience of positive mental health.
Emotional well-being | Change from baseline to four month follow-up (up to 12 months)
  Stress and depression items from modified Depression Anxiety Stress Scales (DASS-21). Participants rate the 14 stress and depression items on a 4-point Likert scale from 0=never to 3 = more than two times. Total scores are calculated for the stress and depression subscales with a range of 0 to 21 with higher scores indicating higher stress or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Crooks, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Graybill, E. C., Varjas, K., Meyers, J., Dever, B. V., Greenberg, D., Roach, A. T., & Morillas, C. (2015). Demographic trends and advocacy experiences of Gay-Straight Alliance advisors. Journal of LGBT Youth, 12(4), 436-461.
- [Background] Heck NC. The Potential to Promote Resilience: Piloting a Minority Stress-Informed, GSA-Based, Mental Health Promotion Program for LGBTQ Youth. Psychol Sex Orientat Gend Divers. 2015 Sep;2(3):225-231. doi: 10.1037/sgd0000110. PMID 26366425
- [Background] Heck, N. C., Flentje, A., & Cochran, B. N. (2011). Offsetting risks: High school gay-straight alliances and lesbian, gay, bisexual, and transgender (LGBT) youth. School Psychology Quarterly, 26(2), 161-174.
- [Background] Ioverno S, Belser AB, Baiocco R, Grossman AH, Russell ST. The Protective Role of Gay-Straight Alliances for Lesbian, Gay, Bisexual, and Questioning Students: A Prospective Analysis. Psychol Sex Orientat Gend Divers. 2016 Dec;3(4):397-406. doi: 10.1037/sgd0000193. PMID 28042585
- [Background] Lapointe, A., & Crooks, C. V. (2018). GSA members' experiences with a structured program to promote well-being. Journal of LGBT Youth. doi: 10.1080/19361653.2018.1479672
- [Background] Lapointe, A., & Crooks, C. V. (in preparation). Supports and strategies suggested by educators to enhance the delivery of a mental health promotion program offered in GSAs. Manuscript in preparation for submission to the Journal of Evaluation and Program Planning.
- [Background] Lapointe, A., Dunlop, C., Crooks, C. V. (2018). Feasibility and fit of a mental health promotion program for LGBTQ+ youth. Manuscript accepted for publication in the Journal of Youth Development.
- [Background] Legislative Assembly of Ontario (2012). Bill 13, (Chapter 5) Statutes of Ontario, 2012: An act to amend the Education Act with respect to bullying and other matters. Toronto, ON: Legislative Assembly of Ontario.
- [Background] Lowry R, Johns MM, Gordon AR, Austin SB, Robin LE, Kann LK. Nonconforming Gender Expression and Associated Mental Distress and Substance Use Among High School Students. JAMA Pediatr. 2018 Nov 1;172(11):1020-1028. doi: 10.1001/jamapediatrics.2018.2140. PMID 30264092
- [Background] Padilla YC, Crisp C, Rew DL. Parental acceptance and illegal drug use among gay, lesbian, and bisexual adolescents: results from a national survey. Soc Work. 2010 Jul;55(3):265-75. doi: 10.1093/sw/55.3.265. PMID 20632661
- [Background] Poteat VP, Heck NC, Yoshikawa H, Calzo JP. Gay-Straight Alliances as settings to discuss health topics: individual and group factors associated with substance use, mental health, and sexual health discussions. Health Educ Res. 2017 Jun 1;32(3):258-268. doi: 10.1093/her/cyx044. PMID 28472258
- [Background] Poteat, V. P., Sinclair, K. O., DiGiovanni, C. D., Koenig, B. W., & Russell, S. T. (2013). Gay-straight alliances are associated with student health: A multischool comparison of LGBTQ and heterosexual youth. Journal of Research on Adolescence, 23(2), 319-330.
- [Background] Russell ST, Fish JN. Mental Health in Lesbian, Gay, Bisexual, and Transgender (LGBT) Youth. Annu Rev Clin Psychol. 2016;12:465-87. doi: 10.1146/annurev-clinpsy-021815-093153. Epub 2016 Jan 14. PMID 26772206
- [Background] Saewyc EM, Konishi C, Rose HA, Homma Y. School-Based Strategies to Reduce Suicidal Ideation, Suicide Attempts, and Discrimination among Sexual Minority and Heterosexual Adolescents in Western Canada. Int J Child Youth Family Stud. 2014 Jan 1;5(1):89-112. doi: 10.18357/ijcyfs.saewyce.512014. PMID 26793284
- [Background] Taylor, C., Meyer, E. J., Peter, T., Ristock, J., Short, D., & Campbell, C. (2016). Gaps between beliefs, perceptions, and practices: The every teacher project on LGBTQ-inclusive education in Canadian schools. Journal of LGBT Youth, 13(1-2), 112-140.
- [Background] Taylor, C., Peter, T., McMinn, T. L., Elliott, T., Beldom, S., Ferry, A., Gross, Z., Paquin, S., & Schachter, K. (2011). Every class in every school: The first national climate survey on homophobia, biphobia, and transphobia in Canadian schools. Toronto, ON: EGALE Canada Human Rights Trust.
- [Background] Toomey RB, Ryan C, Diaz RM, Card NA, Russell ST. Gender-nonconforming lesbian, gay, bisexual, and transgender youth: school victimization and young adult psychosocial adjustment. Dev Psychol. 2010 Nov;46(6):1580-9. doi: 10.1037/a0020705. PMID 20822214
- See also: Project website — https://www.csmh.uwo.ca/research/hrp_for_lgbt2q.html